CLINICAL TRIAL: NCT01018849
Title: Role of Vitamin D in Secondary Prevention of Cardiovascular Events
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Creighton University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 08-15149
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Cardiovascular Disease
Keywords: Vitamin D; Cardiac Catheterization; Cardiovascular event; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (cholecalciferol) (Active Comparator): Subjects receive 150,000 IU of Vitamin D3 every 2 months
  Interventions: Dietary Supplement: Cholecalciferol
- Placebo (Placebo Comparator): Subject will receive a placebo - an exact replica of the Vitamin D3 capsule that does not contain the active ingredient, Vitamin D3
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cholecalciferol — cholecalciferol 150,000 IU by mouth every 2 months for 1 year
  Other Names: Vitamin D3
  Arms: Vitamin D (cholecalciferol)
Dietary Supplement: Placebo — placebo by mouth every 2 months for 1 year
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if Vitamin D supplementation helps prevent recurrent cardiovascular events, such as heart attack or stroke, in patients who have already experienced at least one cardiovascular event. This study will investigate if the addition of 150,000 international units of cholecalciferol (vitamin D3) by mouth every 2 months to a subject's medication regimen will prevent further cardiovascular events.

DETAILED DESCRIPTION:
The purpose of this study is to determine if Vitamin D supplementation helps prevent recurrent cardiovascular events, such as heart attack or stroke, in patients who have already experienced at least one cardiovascular event. This study will investigate if the addition of 150,000 international units of cholecalciferol (vitamin D3) by mouth every 2 months to a subject's medication regimen will prevent further cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of age > 19 years at the time informed consent is signed.
* Subject with a diagnosis of unstable angina (with Thrombolysis in Myocardial Infarction (TIMI) score of greater than or equal to 3) / NSTEMI or STEMI,or documented coronary artery disease defined as at least one coronary artery with > 50% occlusion
* Subject who is able to come back to our clinic for follow up visits for at least 1 year after enrollment.

Exclusion Criteria:

* Subject is on treatment with either phenytoin or phenobarbitol or orlistat (since these medications may cause vitamin D deficiency).
* Subject who needs two or more steroid bursts per year for other co-morbid conditions (since steroids may impair vitamin D metabolism).
* Subject is on an investigational drug, which is a new drug class and not part of standard ACS protocol.
* Subject is taking supplements of vitamin D with doses >400 IU/day.
* Subject has hypersensitivity to vitamin D products.
* Subject has history of systemic lupus erythematosus (since vitamin D deficiency is common in this group27).
* Subject has history of sarcoidosis (since they have hypercalcemia and high levels of vitamin D28)
* Subject has history of renal stones.
* Subject has hypercalcemia, which is defined as serum calcium levels >10.6 mg/dl, at the time of screening.
* Subject has end stage renal disease, defined as either chronic kidney disease stage V or requiring dialysis (since these patients have altered vitamin D and calcium metabolism).
* Subject has systemic disease (including terminal cancer, cirrhosis, end stage COPD etc.,) with reduced (<12 months) life expectancy.
* Subject has a history of psychiatric illness/condition that would interfere with his/her ability to understand or complete the requirements of the study.
* Subject has any condition that in the opinion of the investigator places the subject at an unacceptable risk as a participant in this study.
* Subject is pregnant.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2013-07 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
To give oral vitamin D supplements and raise the blood levels of 25-OH D in the study subjects to >30ng/ml. | 1 year
To see if raising the serum 25(OH) D levels reduces the incidence of cardiovascular events in patients with coronary artery disease (CAD). | 1 year

SECONDARY OUTCOMES:
To see if higher serum 25(OH) D levels will help in better control of blood pressure. | 1 year
To perform proteomics analysis to: a) Extract total protein; b) Profile protein expression in 2-DE and /or 2-DLC and direct mass spectrometric analysis (dMS) on the serum of vitamin D supplemented and placebo subjects. | 1 year
To compare protein expression profiles and/or MS spectrum pattern recognition, and identify differentially expressed proteins in vitamin D supplemented and placebo subjects. | 1 year
To obtain bone mineral density measurements (by DXA) and assess bone markers in subjects with known coronary artery disease | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Laura Armas, MD, Principal Investigator — University of Nebraska
Locations (2):
- United States (2):
  - The Cardiac Center at Creighton University, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska